CLINICAL TRIAL: NCT02029482
Title: Single-center, Double-blind, Placebo-controlled, Randomized, Parallel-group, Up-titration Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Increasing Doses of ACT-128800 in Healthy Male and Female Subjects
Brief Title: Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACT-128800 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AC-058-109
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Safety and Tolerability
Keywords: ACT-128800
MeSH Terms: interventions — ponesimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT-128800 (Experimental): ACT-128800 tablets, once daily for 3 days at each dose level: 10 mg, 20 mg, 40 mg, 60 mg, 80 mg, and 100 mg.
  Interventions: Drug: ACT-128800
- Placebo (Placebo Comparator): Matching placebo tablets, once daily, for 18 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-128800
  Arms: ACT-128800
Drug: Placebo
  Arms: Placebo

SUMMARY:
This was a single-center, randomized, double-blind, placebo-controlled, up-titration Phase 1 study. Sixteen subjects in two groups (at least 40% of subjects of either male or female sex), with 12 subjects in the active treatment group with an up-titration scheme from 10 to 100 mg, and 4 subjects in the placebo treatment group. Subjects were administered ascending doses of ACT-128800/placebo once daily for 3 days at each dose level: 10 mg, 20 mg, 40 mg, 60 mg, 80 mg, and 100 mg.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure.
* Age between 18 and 65 years (inclusive) at screening.
* Body mass index (BMI) between 18 and 30 kg/m^2 (inclusive).
* Women of childbearing potential were required to have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to first drug intake and have agreed to use two methods of contraception from the screening visit until 2 months after study drug discontinuation.
* Systolic blood pressure 100-150 mmHg, diastolic blood pressure 50-90 mmHg measured on the leading arm, and heart rate 50-95 beats per minute (inclusive) measured by electrocardiography (ECG) after 5 minutes in the supine position at screening.
* ECG without clinically relevant abnormalities at screening.
* Hematology and clinical chemistry results not deviating from the normal range to a clinically relevant extent at screening.
* Negative results from urine drug screen at screening.
* Ability to communicate well with the investigator and to understand and comply with the requirements of the study.

Exclusion Criteria:

* ECG recording; PQ/PR interval > 200 ms at screening.
* Pregnant or lactating women.
* Known hypersensitivity to any excipients of the drug formulation.
* Known hypersensitivity to beta2 adrenergic receptor agonists.
* Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access or puncture; veins with a tendency to rupture during or after puncture).
* Treatment with another investigational drug within 3 months prior to screening.
* Excessive caffeine consumption, defined as ≥ 800 mg per day at screening. History or clinical evidence of any disease and/or existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism or excretion of the study drug.
* Smoking within the last month prior to screening.
* Any immunosuppressive treatment within 6 weeks before study drug administration.
* Previous treatment with any prescribed or over-the-counter medications (including herbal medicines such as St John's Wort) within 2 weeks prior to screening or 5 half-lives of the drug, whichever is longer.
* Loss of 250 mL or more of blood within 3 months prior to screening.
* Lymphopenia (< 1,000 cells/μL).
* Viral, fungal, bacterial or protozoal infection within 4 weeks before study drug administration (e.g., active herpes and/or cytomegalovirus infection).
* History or clinical evidence suggestive of active or latent tuberculosis at screening.
* Positive results from the hepatitis serology, except for vaccinated subjects, at screening.
* Positive results from the human immunodeficiency virus serology at screening.
* Forced expiratory volume in 1 second (FEV1) or forced vital capacity (FVC) < 80% of the predicted value, or FEV1/FVC ratio < 0.7 at screening.
* History of asthma or chronic obstructive pulmonary disease.
* Any cardiac condition or illness (including ECG abnormalities) with a potential to increase the cardiac risk of the subject in the standard 12-lead ECG and 24-hour 3-lead Holter ECG at screening.
* History of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Familial history of sick-sinus syndrome.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening. Alcohol abuse is defined as regular weekly intake of more than 21 units.
* Legal incapacity or limited legal capacity at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 18 in systolic blood pressure | 18 days
  Blood pressure was measured using an automatic oscillometric device, always on the leading arm (i.e., leading arm right = writing with right hand).
  Measurements were recorded from the subject in the supine position after having rested for a 5-minute period.
Change from baseline to Day 18 in diastolic blood pressure | 18 days
  Blood pressure was measured using an automatic oscillometric device, always on the leading arm (i.e., leading arm right = writing with right hand).
  Measurements were recorded from the subject in the supine position after having rested for a 5-minute period.
Change from baseline to Day 18 in pulse rate | 18 days
  Pulse rate was measured using an automatic oscillometric device, always on the leading arm (i.e., leading arm right = writing with right hand).
  Measurements were recorded from the subject in the supine position after having rested for a 5-minute period.
Change from baseline to Day 18 in body temperature | 18 days
  Body temperature was measured in the supine position using the same thermometer throughout the study.

SECONDARY OUTCOMES:
Change from baseline to Day 10 in mean absolute lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte counts were determined with standard commercially available assay kits.
Change from baseline to Day 10 in mean T cell (Cluster of differentiation (CD) CD3+) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean B cell (CD3-/CD19+) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean natural killer (NK) cell (CD3-/CD56+) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean natural killer T (NKT) cell (CD3+/CD56+) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean CD4+ T-helper cell (CD3+/CD4+) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean T-cytotoxic cell (CD3+/CD8+) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean CD4+T-naive cell (CD45RA+/chemokine receptor type 7 (CCR7+)) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean CD4+ T-central memory cell (CD45RA-/CCR7+) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean CD4+ T-effector memory cell (CD45RA-/CCR7-) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean CD4+ T-effector cell (CD45RA+/CCR7-) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean CD8+ T-naive cell (CD45RA+/CCR7+) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean CD8+ T-central memory cell (CD45RA-/CCR7+) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean CD8+ T-effector memory cell (CD45RA-/CCR7-) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean CD8+ T-effector cell (CD45RA+/CCR7-) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean T-regulatory cell (CD25+/Forkhead box P3 (Foxp3+)) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean skin-homing T-helper cell (Cutaneous lymphocyte antigen (CLA)+/integrin β7-) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Change from baseline to Day 10 in mean gut-homing T-helper cell (CLA-/integrin β7+) lymphocyte count | 10 days
  For each assessment, 1.5 mL of blood was collected aseptically from the subject in the supine position by venipuncture or via an intravenous. catheter placed in an antecubital vein in the arm in ethylenediaminetetraacetic acid containing tubes. Immediately following collection of the required whole blood volume, the tubes were slowly tilted backwards and forwards (no shaking) to bring the anti-coagulant into solution. The anticoagulated whole blood stored at room temperature (20-25 °C) was preferably stained within 12 hours, at the latest 24 hours, and analyzed within 24 hours. The lymphocyte subset counts were analyzed by fluorescence activated cell sorting.
Maximum plasma concentration (Cmax) of ACT-128800 on Days 9 and 18 | 18 days
  Blood samples for pharmacokinetic analysis were taken following drug administration on study Day 9 (Day 3 of the dosing period with 40 mg) and study Day 18 (Day 3 of the dosing period with 100 mg) and Cmax of ACT-128800 was determined by non-compartmental analysis.
Area under the plasma concentration-time curve from time 0 to 24 hours (AUC0-24) of ACT-128800 on Days 9 and 18 | 18 days
  Blood samples for pharmacokinetic analysis were taken following drug administration on study Day 9 (Day 3 of the dosing period with 40 mg) and study Day 18 (Day 3 of the dosing period with 100 mg) and AUC0-24 of ACT-128800 was determined by non-compartmental analysis.
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-infinity) of ACT-128800 on Day 18 | 18 days
  Blood samples for pharmacokinetic analysis were taken following drug administration on study Day 18 (Day 3 of the dosing period with 100 mg) and AUC0-infinity of ACT-128800 was determined by non-compartmental analysis.
Time to reach maximum plasma concentration (tmax) of ACT-128800 on Days 9 and 18 | 18 days
  Blood samples for pharmacokinetic analysis were taken following drug administration on study Day 9 (Day 3 of the dosing period with 40 mg) and study Day 18 (Day 3 of the dosing period with 100 mg) and tmax of ACT-128800 was determined by non-compartmental analysis.
Terminal half-life (t1/2) of ACT-128800 on Day 18 | 18 days
  Blood samples for pharmacokinetic analysis were taken following drug administration on study Day 18 (Day 3 of the dosing period with 100 mg) and t1/2 of ACT-128800 was determined by non-compartmental analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS, DCPSA, Principal Investigator — Quintiles Drug Research Unit
Locations (1):
- Quintiles Drug Research Unit at Guy's Hospital, London, United Kingdom